CLINICAL TRIAL: NCT02596126
Title: Secondary Prevention of Cardiovascular Disease in the Elderly Trial
Acronym: SECURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Collaborators: Charite University, Berlin, Germany (Other); Centre Hospitalier Universitaire de Besancon (Other); Wroclaw Medical University (Other); Semmelweis University (Other); General University Hospital, Prague (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); London School of Hygiene and Tropical Medicine (Other); Ferrer Internacional S.A. (Industry); Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 633765; 2015-002868-17 (EudraCT Number)
Record Dates: First submitted 2015-10-05; First posted 2015-11-04 (Estimated); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2021-08

CONDITIONS: Myocardial Infarction; Cardiovascular Disease
Keywords: Polypill; Prevention of Secondary Cardiovascular Disease; Cardiovascular Disease; Myocardial Infarction; Cardiovascular Combination Polypill AAR; Cardiovascular Disease in the Elderly; Adherence; SECURE; Elderly; Secondary Cardiovascular Disease; Secondary Cardiovascular Prevention; Randomized Cardiovascular Trial; Randomized Trial; Cardiovascular Polypill
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases | interventions — Platelet Aggregation Inhibitors; Hypolipidemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Prevention for Secondary CV (Active Comparator): Patients allocated to the usual care arm will receive standard of care therapies for secondary prevention according to the ESC guidelines. Drugs and doses will be left at the discretion of the treating physicians..
  Interventions: Drug: Treatment Prevention for Secondary CV
- Cardiovascular Polypill (Experimental): Patients allocated to the experimental arm will receive a cardiovascular polypill containing aspirin 100 mg, atorvastatin (40 or 20 mg) and ramipril (2.5, 5 or 10 mg) taken orally once a day.
  Interventions: Drug: Cardiovascular Polypill

INTERVENTIONS:
Drug: Cardiovascular Polypill — Cardiovascular Polypill contains Aspirin, Atorvastatin and Ramipril.
  Participants will receive one of the following cardiovascular polypill:
  (A) Aspirin 100 mg, Atorvastatin 40mg, and Ramipril (2.5 mg, or 5 mg, or 10mg).
  or
  (B) Aspirin 100 mg, Atorvastatin 20mg, and Ramipril (2.5 mg, or 5 mg, or 10mg).
  Other Names: Polypill
  Arms: Cardiovascular Polypill
Drug: Treatment Prevention for Secondary CV — ESC Guideline (2013 guideline on management of stable coronary disease) recommended pharmacological treatment for event prevention.
  Other Names: Antiplatelet agents; Lipid Lowering Agents; Renin-angiotensin-aldosterone system blockers
  Arms: Treatment Prevention for Secondary CV

SUMMARY:
The purpose of this study is to evaluate the efficacy of a polypill strategy containing aspirin (100 mg), ramipril (2.5, 5 or 10 mgs), and atorvastatin (40 mgs) compared with the standard of care (usual care according to the local clinical practices at each participating country) in secondary prevention of major cardiovascular events (cardiovascular death, nonfatal myocardial infarction, nonfatal ischemic stroke, and urgent revascularization) in elderly patients with a recent myocardial infarction.

DETAILED DESCRIPTION:
A total number of 2499 patients have been randomized (1:1) to treatment arms. Patients will be recruited across seven countries in Europe (Spain, Italy, Germany, France, Hungary, Poland, and Czech Republic).

Patients will be ≥65 years old and diagnosed with a type 1 myocardial infarction within 6 months prior to study enrolment.

Once the inclusion and exclusion criteria are confirmed, patients will be included in the study after signing informed consent.

Randomization will take place within 6 months of the index event (AMI type I) in a 1:1 ratio to one of the two arms:

* Cardiovascular Polypill (containing Aspirin, Ramipril, and Atorvastatin)
* Usual care

Patients will be followed up for a minimum of 2 years and a maximum of 5 years.

There will be 3 follow up visits at month 6, 12 and 24 and telephone follow up calls at month 18, 36, 48 and 60

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with a type 1 myocardial infarction within the previous 6 months.
2. Subjects must be ≥65 years old, presenting with at least one of the following additional conditions:

   * Documented diabetes mellitus or previous treatment with oral hypoglycemic drugs or insulin.
   * Mild to moderate renal dysfunction: creatinine clearance 60-30 mL/min/1.73 m2.
   * Prior myocardial infarction: defined as an AMI occurring before the index event documented in a medical report.
   * Prior coronary revascularization: coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI).
   * Prior stroke: history of a documented stroke, defined as an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of central nervous system tissue, not resulting in death.
   * Age ≥ 75 years.
3. Signing informed consent.

Exclusion Criteria:

1. Unable to sign informed consent.
2. Contraindications to any of the components of the polypill.
3. Living in a nursing home.
4. Mental illness limiting the capacity of self-care.
5. Participating in another clinical trial.
6. Severe congestive heart failure (NYHA III-IV).
7. Severe renal disease (Creatinine Clearance (CrCl) <30ml/min/1.73 m2).
8. Need for oral anticoagulation at the time of randomization or planned in the future months.
9. Any condition limiting life expectancy <2 years, including but not limited to active malignancy.
10. Significant arrhythmias (including unresolved ventricular arrhythmias or atrial fibrillation).
11. Scheduled coronary revascularization (patients can be randomized after final revascularization is completed within the prespecified timeframe).
12. Do not agree to the filing, forwarding and use of his/ her pseudonymised data.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2499 (Actual)
Dates: Start 2016-07; Primary Completion 2021-10-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Principal Investigator — Centro Nacional de Investigaciones Cardiovasculares Carlos III; Jose Maria Castellano Vazquez, MD, PhD, Study Director — Centro Nacional de Investigaciones Cardiovasculares Carlos III
Locations (113):
- Czechia (9):
  - Všeobecná fakultní nemocnice v Praze, Prague, Prague
  - Fakultní nemocnice Královské Vinohrady, Prague, Praha 10
  - Nemocnice Na Homolce, Prague, Praha 5
  - Nemocnice Rudolfa a Stefanie Benešov, Benešov
  - Nemocnice Jihlava, Jihlava
  - Krajská necmonice Liberec, Liberec
  - Fakultní nemocnice Olomouc, Olomouc
  - Nemocnice Slaný, Slaný
  - Nemocnice Podlesí, Třinec
- France (14):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Lyon, Bron
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier Metropole Savoie, Chambéry
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Régional et Universitaire de Lille, Lille
  - Centre Hospitalier St Joseph St Luc, Lyon
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital Bichât, Paris
  - Centre hospitalier Universitaire de Bordeaux, Pessac
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Germany (17):
  - Klinik am See, Rehabilitationszentrum für innere Medizin, Rüdersdorf, Brandenburg
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau, State of Berlin
  - Medical Park Berlin Humboldtmühle, Tegel, State of Berlin
  - Brandenburgklinik Berlin-Brandenburg GmbH, Haus Brandenburg/ Kardiologie, Waldsiedlung, State of Berlin
  - GLG Fachklinik Wolletzsee GmbH, Angermünde
  - AVK Vivantes Rehabilitation GmbH, Berlin
  - DRK- Kliniken Berlin/ Köpenick, Berlin
  - Maria Heimsuchung Caritas-Klinik Pankow, Berlin
  - Jüdisches Krankenhaus, Berlin
  - Charité - Universitätsmedizin Berlin, Centrum für Schlaganfallforschung (CSB), Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - Vivantes Klinikum Spandu, Berlin
  - DRK Klinik Berlin Westend, Berlin
  - GK Havelhöhe, Berlin
  - Gesundheitszentrum Bitterfeld /Wolfen GmbH, Bitterfeld-Wolfen
  - Mediclin Reha-Zentrum Spreewald Fachklinik für innere Medizin, Burg
  - MediClin Herzzentrum Coswig, Coswig
- Hungary (7):
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászati Klinika, Budapest
  - Fővárosi Szent János Kórház, Budapest
  - Szent Rókus Kórház és Intézményei, Budapest
  - Békés Megyei Pándy Kálmán Kórház, Gyula
  - Bács- Kiskun Megyei Kórház, Kecskemét
  - Fejér Megyei Szent György Egyetemi Kórház, Székesfehérvár
  - Sydó és Tsa Kft., Veszprém
- Italy (26):
  - IRCCS Fondazione S. Maugeri Istit. di Cassano Murge, Cassano delle Murge, BA
  - IOB-Policlinico San Marco, Osio Sotto, BG
  - Ospedale Bolognini di Seriate - ASST BERGAMO EST, Seriate, BG
  - ASST di Bergamo Ovest-Ospedale di Treviglio, Treviglio, BG
  - ASST Degli Spedali Civili di Brescia, Brescia, BS
  - Ospedale S.Lazzaro, Alba, CN
  - Ospedale Generale di Zona-Ospedale Valduce, Como, CO
  - ASL FG Ospedale "Teresa Masselli Mascia", San Severo, FG
  - Ospedale Misericordia ASL 9 Grosseto, Grosseto, GR
  - Ospedale Sacro Cuore di Gesù, Gallipoli, LE
  - ASST Di Monza-Presidio Ospedaliero di Desio, Desio, MB
  - ASST Di Monza-Ospedale San Gerardo, Monza, MB
  - IRCCS Ospedale Policlinico di Milano, Milan, MI
  - Centro Cardiologico Monzino SpA, Milan, MI
  - ASST Santi Paolo e Carlo-Ospedale San Paolo-Polo Univ., Milan, MI
  - IRCCS-Fondazione Don Carlo Gnocchi, Milan, MI
  - IRCCS Istituto Clinico Humanitas, Rozzano, MI
  - IRCCS Policlinico San Donato, San Donato Milanese, MI
  - Ospedale di Sassuolo S.P.A., Sassuolo, MO
  - ASST Rhodense Ospedale di Passirana, Passirana, Passirana-rho
  - Presidio Ospedaliero San Filippo Neri-ASL Roma E, Roma, RM
  - A.O. San Camillo Forlanini, Roma, RO
  - Ospedale Ss Giovanni di Dio e Ruggi d'Aragona, Salerno, SA
  - Casa di Cura Villa Bianca, Trento, TN
  - AAS3 "Alto Friuli, Collinare, Medio Friuli" Ospedale di San Daniele del Friuli-Tolmezzo sede di S. D. del Friuli, San Daniele del Friuli, UD
  - ASST Della Valle Olona-Ospedale di Saronno, Saronno, VA
- Poland (10):
  - Samodzielny Publiczny Szpital Kliniczny nr 7, Śląskiego Uniwersytetu Medycznego w Katowicach, Górnośląskie Centrum Medyczne im. prof. Leszka Gieca, Katowice, Ochojec
  - Uniwersyteckie Centrum Kliniczn, Gdansk
  - Szpital Wielospecjalistyczny im. Dr. Ludwika Błażka w Inowrocławiu, Inowrocław
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - Zespół Opieki Zdrowotnej w Kłodzku, Kłodzko
  - Wojewódzki Szpital Specjalistyczny w Legnicy, Legnica
  - Samodzielny Publiczny Zespół Opieki Zdrowotnej w Świdnicy, Swidnica
  - Specjalistyczny Szpital im. Dra Alfreda Sokołowskiego, Wałbrzych
  - Centrum Kardiologiczne "Pro Corde" Sp. z o.o., Wroclaw
  - Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ, Wroclaw
- Spain (30):
  - Hospital Univeristari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - H.C.U.de Santiago De Compostela, Santiago de Compostela, Galicia
  - Complejo Asistencial Universitario de Leon, León, Leon
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital General de Villalba, Collado Villalba, Madrid
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario QuironSalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Infanta Elena, Valdemoro, Madrid
  - H.C.U. Virgen De La Arrixaca De Murcia, El Palmar, Murcia
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall D'hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia de Cordoba, Córdoba
  - Hospital La Luz Quiron, Madrid
  - C.H.U. Ruber Juan Bravo, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinic Universitari de Valencia, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia

REFERENCES:
- [Derived] Castellano JM, Pocock SJ, Bhatt DL, Quesada AJ, Owen R, Fernandez-Ortiz A, Sanchez PL, Marin Ortuno F, Vazquez Rodriguez JM, Domingo-Fernandez A, Lozano I, Roncaglioni MC, Baviera M, Foresta A, Ojeda-Fernandez L, Colivicchi F, Di Fusco SA, Doehner W, Meyer A, Schiele F, Ecarnot F, Linhart A, Lubanda JC, Barczi G, Merkely B, Ponikowski P, Kasprzak M, Fernandez Alvira JM, Andres V, Bueno H, Collier T, Van de Werf F, Perel P, Rodriguez-Manero M, Alonso Garcia A, Proietti M, Schoos MM, Simon T, Fernandez Ferro J, Lopez N, Beghi E, Bejot Y, Vivas D, Cordero A, Ibanez B, Fuster V; SECURE Investigators. Polypill Strategy in Secondary Cardiovascular Prevention. N Engl J Med. 2022 Sep 15;387(11):967-977. doi: 10.1056/NEJMoa2208275. Epub 2022 Aug 26. PMID 36018037
- [Derived] Buttgereit T, Palmowski A, Forsat N, Boers M, Witham MD, Rodondi N, Moutzouri E, Navidad AJQ, Van't Hof AWJ, van der Worp B, Coll-Planas L, Voshaar M, de Wit M, da Silva J, Stegemann S, Bijlsma JW, Koeller M, Mooijaart S, Kearney PM, Buttgereit F. Barriers and potential solutions in the recruitment and retention of older patients in clinical trials-lessons learned from six large multicentre randomized controlled trials. Age Ageing. 2021 Nov 10;50(6):1988-1996. doi: 10.1093/ageing/afab147. PMID 34324628

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited across seven countries in Europe (Spain, Italy, Germany, France, Hungary, Poland, and Czech Republic). Patients were ≥65 years old and diagnosed with a type 1 myocardial infarction within 6 months prior to study enrolment.
Pre-assignment Details: Patients can be screened at any time within the first 8 weeks after index event (type 1 myocardial infarction) whenever they are clinically stable and ready to receive secondary prevention therapy, including the hospital phase. Patients with ventricular arrhythmias needing further evaluation of therapy.
Groups:
- Cardiovascular Polypill: Patients allocated to the experimental arm will receive a cardiovascular polypill containing aspirin 100 mg, atorvastatin (40 or 20 mg) and ramipril (2.5, 5 or 10 mg) taken orally once a day.
  Cardiovascular Polypill: Cardiovascular Polypill contains Aspirin, Atorvastatin and Ramipril.
  Participants will receive one of the following cardiovascular polypill:
  (A) Aspirin 100 mg, Atorvastatin 40mg, and Ramipril (2.5 mg, or 5 mg, or 10mg).
  or
  (B) Aspirin 100 mg, Atorvastatin 20mg, and Ramipril (2.5 mg, or 5 mg, or 10mg).
Period: Overall Study
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Started | 1241 | 1258
Completed | 1222 | 1228
Not Completed | 19 | 30
Not completed — Lost to Follow-up | 12 | 21
Not completed — Protocol Violation | 7 | 9

BASELINE CHARACTERISTICS:
Population: A total of 2499 participants (Treatment Prevention for Secondary CV - 1241; Cardiovascular Polypill - 1258) were included in the study. A total of 33 (Treatment Prevention for Secondary CV - 12; Cardiovascular Polypill - 21) participants were lost to follow-up as described in the "Results Participant Flow". The results were presented for a total of 1229 participants in the "Treatment Prevention for Secondary CV" and 1237 participants in the "Cardiovascular Polypill".
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill | Total
Number analyzed (Participants) | 1229 | 1237 | 2466
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1229 | 1237 | 2466
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 381 | 384 | 765
  Male | 848 | 853 | 1701
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 1211 | 1221 | 2432
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 13 | 31
Region of Enrollment [Number; unit: participants]
  Hungary | 45 | 45 | 90
  Czechia | 87 | 85 | 172
  Poland | 60 | 63 | 123
  Italy | 365 | 366 | 731
  France | 70 | 74 | 144
  Germany | 184 | 182 | 366
  Spain | 418 | 422 | 840

OUTCOME MEASURES:

1. Primary Outcome: Major Cardiovascular Adverse Events (MACE)
Description: The incidence of the first occurrence of any component of the following composite endpoint, as adjudicated by the Clinical Events Committee:
  * Cardiovascular death.
  * Any nonfatal type 1 myocardial infarction.
  * Any nonfatal ischemic stroke.
  * Any urgent coronary revascularization not resulting in death.
Time Frame: Up to 5 years
Measure: Number; unit: number of adjudicated events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of adjudicated events | 156 | 118
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Non-Inferiority — Non-inferiority hypothesis will be tested using a univariable Cox PH regression model including treatment group as the only covariate and stratified by country. One-sided non-inferiority test on the primary endpoint where the alpha level will be set to 2.5%. All statistical analyses will use 95% confidence intervals (CI). If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a log-rank test; p < 0.025, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.6 to 0.96]
Statistical Analysis 2: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Superiority — If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a logrank test; p < 0.05, Log Rank

2. Secondary Outcome: Efficacy Endpoints
Description: Treatment adherence at 6 months measured using the Morisky-Medication Adherence Scale (8 item) Questionnaire (MMAS-8). Results: Low adherence (0-5); Medium adherence (6-7) and High adherence (8). The number and percentage of patients with low (0-5), medium (6-7) and high (8) adherence will be reported by treatment group.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
percentage of participants
  Low adherence (0-5) | 9.5 | 5.5
  Medium adherence (6-7) | 27.8 | 24.0
  High adherence (8) | 62.7 | 70.6
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - Treatment adherence at 6 months; Test type: Equivalence — Treatment adherence is measured at visit 1 (6 months) and visit 3 (24 months) using the Morisky-Medication Adherence Scale (8 item) Questionnaire (MMAS-8). The number and percentage of patients with low (0-5), medium (6-7) and high (8) adherence will be reported by treatment group. The distributions of the MMAS-8 score at 6 months and 24 months will be compared between treatment groups using an ordinal logistic regression model; p < 0.005, Chi-squared; Risk Ratio (RR) = 1.13, 95% CI 2-sided [1.06 to 1.2]

3. Secondary Outcome: Safety Endpoints
Description: All-cause mortality.
Time Frame: Up to 5 Years
Measure: Number; unit: number of events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of events | 117 | 115
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - All-cause death; Test type: Superiority — Time to first event will be investigated using Cox proportional hazards regression. Hazard ratios and 95% confidence intervals will be obtained from the Cox proportional hazards model. P-values will be obtained using the log-rank test; p < 0.05, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.75 to 1.25]

4. Secondary Outcome: Efficacy Endpoints
Description: Treatment adherence at 24 months measured using the Morisky-Medication Adherence Scale (8 item) Questionnaire (MMAS-8). Results: Low adherence (0-5); Medium adherence (6-7) and High adherence (8). The number and percentage of patients with low (0-5), medium (6-7) and high (8) adherence will be reported by treatment group.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
percentage of participants
  Low adherence (0-5) | 6.9 | 4.2
  Medium adherence (6-7) | 29.8 | 21.7
  High adherence (8) | 63.2 | 74.1
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - Treatment adherence at 24 months; Test type: Equivalence — Treatment adherence is measured at visit 1 (6 months) and visit 3 (24 months) using the Morisky- Medication Adherence Scale (8 item) Questionnaire (MMAS-8). The number and percentage of patients with low (0-5), medium (6-7) and high(8) adherence will be reported by treatment group. The distributions of the MMAS-8 score at 6 months and 24 months will be compared between treatment groups using an ordinal logistic regression model; p < 0.005, Chi-squared; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [1.1 to 1.25]

5. Secondary Outcome: Efficacy Endpoints
Description: The systolic Blood Pressure measured in millimeters of mercury (mmHg) at visit 1 (6 months). Mean and standard deviation will be reported by treatment group.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
millimeters of mercury (mmHg) | 134.8 (18.1) | 134.4 (17.7)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - SBP - 6 months; Test type: Equivalence — The following three CV risk factors, systolic blood pressure(SBP), diastolic blood pressure (DBP) and low-density lipoprotein (LDL) cholesterol levels are measured at baseline, visit 1 (6 months), visit 2 (12 months) and visit 3 (24 months).For each of the three risk factors the frequency, mean and standard deviation at each visit will be reported by treatment group. The difference in mean change from baseline between groups will be compared using ANCOVA; p < 0.05, ANCOVA — The difference in mean change from baseline between groups will be compared using ANCOVA (adjusting for baseline levels) at 6 months, 12 months and 24 months. The difference in mean change adjusting for baseline and 95% CI will be reported; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.8 to 1.2]

6. Secondary Outcome: Efficacy Endpoints
Description: The systolic Blood Pressure measured in millimeters of mercury (mmHg) at visit 2 (12 months). Mean and standard deviation will be reported by treatment group.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
millimeters of mercury (mmHg) | 135.0 (18.0) | 136.3 (17.5)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - SBP - 12 months; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.05, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-0.1 to 3]

7. Secondary Outcome: Efficacy Endpoints
Description: The systolic Blood Pressure measured in millimeters of mercury (mmHg) at visit 3 (24 months). Mean and standard deviation will be reported by treatment group.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
millimeters of mercury (mmHg) | 135.5 (17.1) | 135.2 (16.9)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - SBP - 24 months; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.05, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.7 to 1.4]

8. Secondary Outcome: Efficacy Endpoints
Description: The Diastolic Blood Pressure measured in millimeters of mercury (mmHg) at visit 1 (6 months). Mean and standard deviation will be reported by treatment group. The frequency, mean and standard deviation at each visit will be reported by treatment group.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
millimeters of mercury (mmHg) | 74.2 (9.9) | 74.3 (10.2)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - DBP - 6 months; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.05, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.7 to 1]

9. Secondary Outcome: Efficacy Endpoints
Description: The Diastolic Blood Pressure measured in millimeters of mercury (mmHg) at visit 2 (12 months). Mean and standard deviation will be reported by treatment group. The frequency, mean and standard deviation at each visit will be reported by treatment group.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
millimeters of mercury (mmHg) | 74.1 (9.8) | 74.7 (9.9)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - DBP - 12 months; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.05, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.1 to 1.6]

10. Secondary Outcome: Efficacy Endpoints
Description: The Diastolic Blood Pressure measured in millimeters of mercury (mmHg) at visit 3 (24 months). Mean and standard deviation will be reported by treatment group. The frequency, mean and standard deviation at each visit will be reported by treatment group.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
millimeters of mercury (mmHg) | 74.9 (9.7) | 74.8 (10.1)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - DBP - 24 months; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.05, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.9 to 1]

11. Secondary Outcome: Efficacy Endpoints
Description: Low-density lipoprotein (LDL) cholesterol levels measured in mg/dL at visit 2 (12 months). Mean and standard deviation will be reported by treatment group. The frequency, mean and standard deviation at each visit will be reported by treatment group.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
mg/dL | 66.3 (25.4) | 69.2 (24.7)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - LDL cholesterol - 12 months; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.05, ANCOVA; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-0.2 to 4.4]

12. Secondary Outcome: Efficacy Endpoints
Description: Low-density lipoprotein (LDL) cholesterol levels measured in mg/dL at visit 3 (24 months). Mean and standard deviation will be reported by treatment group. The frequency, mean and standard deviation at each visit will be reported by treatment group.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
mg/dL | 67.2 (25.4) | 67.7 (23.6)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - LDL cholesterol - 24 months; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p < 0.05, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.5 to 2.4]

13. Secondary Outcome: Efficacy Endpoints
Description: The incidence of the first occurrence of any component of the following composite endpoint, as adjudicated by the Clinical Events Committee: Cardiovascular death (CV death); Acute Myocardial Infarction (MI) type 1; stroke. Measured in number of cases.
Time Frame: Up to 5 years
Measure: Number; unit: number of events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of events | 144 | 101
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Non-Inferiority — Non-inferiority hypothesis will be tested using a univariable Cox PH regression model including treatment group as the only covariate and stratified by country. One-sided non-inferiority test on the primary endpoint where the alpha level will be set to 2.5%. All statistical analyses will use 95% confidence intervals (CI).If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a log-rank test; p < 0.025, Regression, Cox; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.54 to 0.90]
Statistical Analysis 2: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Superiority — If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a logrank test; p < 0.05, Log Rank

14. Secondary Outcome: Efficacy Endpoints
Description: The incidence of the first occurrence of the Cardiovascular (CV) death. Measured in number of cases.
Time Frame: Up to 5 years
Measure: Number; unit: number of events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of events | 71 | 48
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; p < 0.025, Regression, Cox; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.47 to 0.97]
Statistical Analysis 2: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Superiority — If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a logrank test; p < 0.05, Log Rank

15. Secondary Outcome: Efficacy Endpoints
Description: The incidence of the first occurrence of of the Nonfatal type 1 myocardial infarction. Measured in number of cases.
Time Frame: Up to 5 years
Measure: Number; unit: number of events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of events | 62 | 44
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; p < 0.025, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.48 to 1.05]
Statistical Analysis 2: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Superiority — If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a logrank test; p < 0.05, Log Rank

16. Secondary Outcome: Efficacy Endpoints
Description: The incidence of the first occurrence of the Nonfatal ischemic stroke. Measured in number of cases.
Time Frame: Up to 5 years
Measure: Number; unit: number of events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of events | 27 | 19
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; p < 0.025, Regression, Cox; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.39 to 1.26]
Statistical Analysis 2: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Superiority — If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a logrank test; p < 0.05, Log Rank

17. Secondary Outcome: Efficacy Endpoints
Description: The incidence of the first occurrence of the Urgent coronary revascularization. Measured in number of cases.
Time Frame: Up to 5 years
Measure: Number; unit: number of events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of events | 28 | 27
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; p < 0.025, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.57 to 1.63]
Statistical Analysis 2: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Test type: Superiority — If the non-inferiority hypothesis is confirmed, it will be followed with a test of superiority using a logrank test; p < 0.05, Log Rank

18. Secondary Outcome: Efficacy Endpoints
Description: Domain "effectiveness" of the Patient satisfaction measured at visit 1 (6 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM (version 1.4) has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain (effectiveness) the response was measured on a Likert-type scale of 5 or 7 points. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction (higher scores reflect higher patient satisfaction with medication).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 69.17 (17.57) | 72.26 (17.85)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Patient satisfaction is measured at visit 1 (6 months) and visit 3 (2 years) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument comprising of four domains: effectiveness (questions 1 to 3), side effects (questions 4 to 8), convenience (questions 9 to 11) and global satisfaction (questions 12 to 14); Test type: Equivalence — Mean and standard devation for each score will be reported by treatment group at 6 months and 2 years. Comparison of mean scores between treatment groups at 6 months and 2 years will be made using a two-sample t-test. The difference in mean score and 95% CI will be reported; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 3.09, 95% CI 2-sided [1.38 to 4.79]

19. Secondary Outcome: Efficacy Endpoints
Description: Domain "Side effects score" of the Patient satisfaction measured at visit 1 (6 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain the response was on a Likert-type scale of 5 or 7 points, except for question 4 which a yes/no question about the presence of side effects is asked. If the answer to this question is no (no side effects reported by the participant), other questions will not be asked (questions 5 to 8), and the total score is automatically computed as the maximum of 100. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 66.71 (23.38) | 61.52 (23.18)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — [test comment as in outcome 18, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -5.19, 95% CI 2-sided [-12.73 to 2.35]

20. Secondary Outcome: Efficacy Endpoints
Description: Domain "Convenience score" of the Patient satisfaction measured at visit 1 (6 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM (version 1.4) has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain (Convenience score) the response was measured on a Likert-type scale of 5 or 7 points. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction (higher scores reflect higher patient satisfaction with medication).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 69.47 (16.87) | 76.56 (14.78)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — [test comment as in outcome 18, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 7.09, 95% CI 2-sided [5.57 to 8.62]

21. Secondary Outcome: Efficacy Endpoints
Description: Domain "Global satisfaction score" of the Patient satisfaction measured at visit 1 (6 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM (version 1.4) has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain (Global satisfaction score) the response was measured on a Likert-type scale of 5 or 7 points. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction (higher scores reflect higher patient satisfaction with medication).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 67.71 (18.53) | 71.50 (18.06)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — [test comment as in outcome 18, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 3.79, 95% CI 2-sided [2.04 to 5.55]

22. Secondary Outcome: Efficacy Endpoints
Description: Domain "effectiveness" of the Patient satisfaction measured at visit 3 (24 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM (version 1.4) has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain (effectiveness) the response was measured on a Likert-type scale of 5 or 7 points. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction (higher scores reflect higher patient satisfaction with medication).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 68.79 (17.65) | 74.06 (17.86)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — [test comment as in outcome 18, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 5.26, 95% CI 2-sided [3.59 to 6.94]

23. Secondary Outcome: Efficacy Endpoints
Description: Domain "Side effects score" of the Patient satisfaction measured at visit 3 (24 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain (Side effects score) the response was on a Likert-type scale of 5 or 7 points, except for question 4 which a yes/no question about the presence of side effects is asked. If the answer to this question is no (no side effects reported by the participant), other questions will not be asked (questions 5 to 8), and the total score is automatically computed as the maximum of 100. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 64.20 (23.14) | 68.75 (24.83)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — [test comment as in outcome 18, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 4.55, 95% CI 2-sided [-4.35 to 13.46]

24. Secondary Outcome: Efficacy Endpoints
Description: Domain "Convenience score" of the Patient satisfaction measured at visit 3 (24 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM (version 1.4) has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain (Convenience score) the response was measured on a Likert-type scale of 5 or 7 points. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction (higher scores reflect higher patient satisfaction with medication).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 70.19 (17.06) | 77.30 (15.95)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — [test comment as in outcome 18, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 7.11, 95% CI 2-sided [5.55 to 8.67]

25. Secondary Outcome: Efficacy Endpoints
Description: Domain "Global satisfaction score" of the Patient satisfaction measured at visit 3 (24 months) using the Treatment Satisfaction Questionnaire for Medication (TSQM) version 1.4 a 14-item psychometric instrument. The TSQM (version 1.4) has 14 questions divided into 4 domains: effectiveness (items 1 to 3), side effects (items 4 to 8), convenience (items 9 to 11), and global satisfaction (items 12 to 14). In this domain (Global satisfaction score) the response was measured on a Likert-type scale of 5 or 7 points. The score is computed by summing the individual TSQM items and then transforming the composite score into a value ranging from 0 to 100, with 0 indicating complete dissatisfaction and 100 indicating complete satisfaction (higher scores reflect higher patient satisfaction with medication).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1229 | 1237
score on a scale | 67.76 (17.87) | 74.36 (17.52)
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; [analysis description as in outcome 18, analysis 1]; Test type: Equivalence — [test comment as in outcome 18, analysis 1]; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 6.60, 95% CI 2-sided [4.93 to 8.27]

26. Secondary Outcome: Safety Endpoints
Description: The incidence of the first occurrence of the Non-cardiovascular death. Measured in number of cases.
Time Frame: Up to 5 Years
Measure: Number; unit: number of events
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
Number analyzed (Participants) | 1241 | 1258
number of events | 46 | 67
Statistical Analysis 1: Comparison: Treatment Prevention for Secondary CV vs Cardiovascular Polypill; Statistical analysis title - Non-cardiovascular death; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.05, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.97 to 2.07]

ADVERSE EVENTS:
Time Frame: Up to 5 Years.
Description: Aspirin, Atorvastatin, and Ramipril have been extensively studied in Phase 1 through Phase 4 clinical studies and their overall safety profile has been well characterized. Thus, appropriate information concerning adverse events were systematically collected and submitted to regulatory authorities
Arm/Group | Treatment Prevention for Secondary CV | Cardiovascular Polypill
All-Cause Mortality (participants affected / at risk) | 117/1229 | 115/1237
Serious Adverse Events (participants affected / at risk) | 220/1229 | 248/1237
Other Adverse Events (participants affected / at risk) | 388/1229 | 404/1237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Prevention for Secondary CV (N=1229) | Cardiovascular Polypill (N=1237)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
abscess (Infections and infestations) | 0 (0) | 1 (1)
abscess drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (2)
acute heart failure (Cardiac disorders) | 1 (1) | 0 (0)
acute kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 9 (9) | 9 (9)
acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
adverse drug reaction (General disorders) | 1 (1) | 0 (0)
allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
anaemia (Blood and lymphatic system disorders) | 9 (10) | 10 (10)
angina pectoris (Cardiac disorders) | 2 (3) | 3 (3)
angina unstable (Cardiac disorders) | 2 (2) | 1 (1)
angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
asthenia (General disorders) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
bacteraemia (Infections and infestations) | 2 (3) | 2 (2)
benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
biliary obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 4 (4) | 2 (2)
bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
cardiac failure (Cardiac disorders) | 1 (2) | 8 (9)
cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
cerebral circulatory failure (Nervous system disorders) | 0 (0) | 1 (1)
cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
chest pain (General disorders) | 15 (16) | 10 (11)
cholangitis (Hepatobiliary disorders) | 0 (0) | 3 (4)
cholangitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 2 (2)
cholelithiasis (Hepatobiliary disorders) | 3 (3) | 2 (3)
cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7)
colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
colitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
complicated fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
confusional state (Nervous system disorders) | 2 (2) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
covid-19 (Infections and infestations) | 5 (5) | 9 (9)
covid-19 pneumonia (Infections and infestations) | 10 (11) | 11 (11)
craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
dementia of the alzheimer's type, with depressed mood (Nervous system disorders) | 0 (0) | 1 (1)
dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dermo-hypodermitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
device dislocation (Product Issues) | 0 (0) | 1 (1)
device related infection (Infections and infestations) | 0 (0) | 1 (1)
diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
diabetic complication(hlgt) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (3)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
dressler's syndrome (Immune system disorders) | 1 (1) | 0 (0)
drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
endocarditis (Infections and infestations) | 1 (1) | 1 (1)
endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
erysipelas (Infections and infestations) | 1 (1) | 0 (0)
escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2)
extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
faecalith (Gastrointestinal disorders) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (5) | 8 (8)
gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal vascular occlusion and infarction (hlt) (Gastrointestinal disorders) | 1 (1) | 0 (0)
general physical health deterioration (General disorders) | 3 (3) | 1 (1)
genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
haematochezia (Gastrointestinal disorders) | 2 (2) | 1 (1)
haematoma (Vascular disorders) | 0 (0) | 2 (2)
haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
haematoma muscle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
haematuria (Renal and urinary disorders) | 7 (9) | 4 (4)
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
haemorrhoids (Vascular disorders) | 1 (1) | 0 (0)
hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
heart failure (Cardiac disorders) | 0 (0) | 1 (1)
hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 4 (5) | 5 (5)
hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
incarcerated parastomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 2 (2) | 1 (1)
injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
interventional procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
intestinal obstruction (Gastrointestinal disorders) | 6 (6) | 0 (0)
iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 3 (3)
lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
malaise (General disorders) | 0 (0) | 1 (1)
malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
mesenteric ischemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 3 (3) | 6 (6)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
open reduction of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pain (General disorders) | 1 (1) | 0 (0)
palliative care (Surgical and medical procedures) | 0 (0) | 1 (1)
palpitations (Cardiac disorders) | 0 (0) | 1 (1)
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 1 (1)
papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
paralysis (Nervous system disorders) | 1 (1) | 0 (0)
partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 17 (17) | 14 (15)
pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
presyncope (Nervous system disorders) | 0 (0) | 1 (1)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
prostatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
prostatitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
psychomotor disadaptation syndrome (Nervous system disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
pyrexia (General disorders) | 2 (3) | 1 (1)
radical cystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4)
renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 0 (0) | 4 (4)
renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
sciatica (Nervous system disorders) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 2 (2)
sepsis (Infections and infestations) | 2 (2) | 2 (2)
septic shock (Infections and infestations) | 1 (1) | 1 (1)
serratia infection (Infections and infestations) | 0 (0) | 1 (1)
shunt infection (Infections and infestations) | 0 (0) | 1 (1)
sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
staphylococcal mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
strangulated hernia (General disorders) | 0 (0) | 1 (1)
streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 3 (3)
subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
sudden death (General disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 7 (9) | 2 (2)
systemic candida (Infections and infestations) | 0 (0) | 1 (1)
temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
terminal state (General disorders) | 0 (0) | 1 (1)
testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
toe amputation (Surgical and medical procedures) | 2 (2) | 0 (0)
tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
torsade de pointe (Cardiac disorders) | 0 (0) | 1 (1)
tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
transurethral bladder resection (Surgical and medical procedures) | 1 (1) | 0 (0)
traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
urethral calculus removal (Surgical and medical procedures) | 1 (1) | 0 (0)
urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
urinary tract infection (Infections and infestations) | 9 (9) | 6 (6)
urosepsis (Infections and infestations) | 1 (1) | 1 (1)
ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
viral infection (Infections and infestations) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Prevention for Secondary CV (N=1229) | Cardiovascular Polypill (N=1237)
Anaemia (Blood and lymphatic system disorders) | 13 (14) | 12 (13)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 9 (11) | 8 (8)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 19 (20) | 16 (19)
Atrial flutter (Cardiac disorders) | 3 (3) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 4 (4)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 4 (4) | 7 (8)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 5 (5)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Blindness transient (Eye disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 7 (7)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 11 (12)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 4 (4) | 4 (4)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Pancreatic failure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pelvic floor dysfunction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (3)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 2 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7) | 4 (4)
Adverse event (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 5 (5)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 28 (31) | 16 (20)
Discomfort (General disorders) | 2 (2) | 0 (0)
Drug intolerance (General disorders) | 2 (3) | 4 (4)
Drug therapeutic incompatibility (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (3) | 0 (0)
Oedema (General disorders) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 12 (12) | 13 (13)
Pacemaker generated arrhythmia (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Stenosis (General disorders) | 1 (1) | 0 (0)
Biloma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Granulomatous liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal fungal infection (Infections and infestations) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (7) | 3 (3)
COVID-19 (Infections and infestations) | 9 (9) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5) | 5 (5)
Respiratory tract infection (Infections and infestations) | 9 (10) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 12 (12) | 10 (13)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Discontinued product administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 9 (9) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angiocardiogram (Investigations) | 1 (1) | 0 (0)
Angiogram (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Biopsy breast (Investigations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 7 (8)
Blood creatinine increased (Investigations) | 1 (2) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure abnormal (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Bronchoscopy (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax (Investigations) | 0 (0) | 1 (1)
Cystoscopy (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Endoscopy gastrointestinal (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Muscle enzyme increased (Investigations) | 0 (0) | 1 (1)
Occult blood (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Renal function test abnormal (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 4 (4) | 4 (4)
Weight decreased (Investigations) | 1 (2) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 10 (10) | 9 (9)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (28) | 14 (15)
Myopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder cancer (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 9 (10) | 13 (13)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 4 (5) | 3 (3)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 15 (17) | 8 (9)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 3 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 5 (7)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 6 (6) | 3 (3)
Renal impairment (Renal and urinary disorders) | 7 (10) | 7 (8)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bendopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (46) | 49 (49)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 17 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 13 (13)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 2 (2) | 2 (2)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carpal tunnel decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 2 (2) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 0 (0) | 1 (2)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Glaucoma surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 2 (2) | 2 (2)
Intra-ocular injection (Surgical and medical procedures) | 0 (0) | 3 (5)
Lymphadenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical counselling (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Pulmonary resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Radiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (2) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 1 (2)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 0 (0) | 2 (2)
Transfusion (Surgical and medical procedures) | 2 (6) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 2 (2)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 2 (2) | 1 (1)
Haemorrhage (Vascular disorders) | 5 (5) | 3 (3)
Haemorrhoids (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 20 (22) | 22 (25)
Hypertensive crisis (Vascular disorders) | 1 (1) | 3 (4)
Hypotension (Vascular disorders) | 15 (15) | 26 (26)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02596126/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT02596126/SAP_001.pdf
  • Informed Consent Form (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02596126/ICF_002.pdf